CLINICAL TRIAL: NCT04232280
Title: A Phase 2, Randomized, Observer-Blind, Placebo-Controlled, Dose-Finding Trial to Evaluate the Safety and Immunogenicity of Cytomegalovirus Vaccine mRNA-1647 in Healthy Adults
Brief Title: Dose-Finding Trial to Evaluate the Safety and Immunogenicity of Cytomegalovirus (CMV) Vaccine mRNA-1647 in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1647-P202
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Cytomegalovirus Infection
Keywords: Moderna; mRNA-1647; Cytomegalovirus; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Congenital; Virus Diseases; Infection Viral; DNA Virus Infections; Messenger RNA
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases; DNA Virus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Observer-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1647 Dose Level A (Experimental): Participants will receive mRNA-1647 vaccine at Dose Level A by intramuscular (IM) injection on Day 1, Day 56, and Day 168.
  Interventions: Biological: mRNA-1647
- mRNA-1647 Dose Level B (Experimental): Participants will receive mRNA-1647 vaccine at Dose Level B by IM injection on Day 1, Day 56, and Day 168.
  Interventions: Biological: mRNA-1647
- mRNA-1647 Dose Level C (Experimental): Participants will receive mRNA-1647 vaccine at Dose Level C by IM injection on Day 1, Day 56, and Day 168.
  Interventions: Biological: mRNA-1647
- Placebo (Placebo Comparator): Participants will receive placebo matching to the mRNA-1647 vaccine dose by IM injection on Day 1, Day 56, and Day 168.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Lyophilized product that is reconstituted with saline then diluted with a special diluent to reach the desired concentration
  Arms: mRNA-1647 Dose Level A; mRNA-1647 Dose Level B; mRNA-1647 Dose Level C
Other: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety and immunogenicity of 3 dose levels of mRNA-1647 cytomegalovirus vaccine in CMV-seronegative and CMV-seropositive healthy adults 18-40 years of age.

DETAILED DESCRIPTION:
mRNA-1647-P202 is a 2-part study. Part 1 of the study evaluates the safety and immunogenicity of 3 dose levels of mRNA-1647 vaccine or placebo, administered on a 0, 2, 6-month schedule in healthy CMV-seronegative and CMV-seropositive males and females, 18 to 40 years of age. A planned interim analysis of safety and immunogenicity through Month 3 (1 month after the second dose) of Part 1 of the study informed the selection of the middle dose level for further development. Part 2 of the study is designed to further evaluate the safety and immunogenicity of the middle dose level of mRNA-1647 vaccine or placebo on a 0, 2, 6-month schedule in approximately 200 healthy participants 18 to 40 years of age, comprised of CMV-seronegative and CMV-seropositive female population, which includes the target population for the pivotal Phase 3 efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-40 years of age (Part 1); Female 18-40 years of age (Part 2)
* Understands and agrees to comply with the trial procedures and provides written informed consent
* According to the assessment of the Investigator, is in good general health and is capable of complying with trial procedures
* Body mass index (BMI) 18-35 kilograms/meter (kg/m^2)
* Female participants must either be of non-childbearing potential or use acceptable methods of contraception from at least 28 days prior to the first vaccination and through 3 months following last vaccination and is not breastfeeding.
* Male participants must agree to practice adequate contraception from the time of the first vaccination and through 3 months after the last vaccination.

Exclusion Criteria:

* Acutely ill or febrile on the day of the first vaccination
* Prior receipt of any CMV vaccine
* Abnormal screening safety laboratory test results
* Diagnosis or condition that, in the judgment of Investigator, is clinically unstable or may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to trial procedures
* Has received or plans to receive a vaccine ≤28 days prior to the first vaccination or plans to receive a non-study vaccine within 28 days prior to or after any study vaccination, except for any licensed influenza vaccine which can be administered >14 days before or after any study vaccination. COVID-19 vaccines (regardless of manufacturer) may be administered >7 days but preferably >14 days before or after any study vaccination, with the intention of prioritizing COVID-19 vaccination over all other considerations.
* Prior receipt of chronic systemic immunosuppressants or immune-modifying drugs
* Receipt of intravenous immunoglobulins or plasma products within 3 months prior to the day of the first study vaccination
* Previous receipt of medications in lipid nanoparticle (LNP) formulation (Part 1 participants only)
* Has donated ≥450 milliliters (mL) of blood products within 28 days of the Screening visit
* Participated in an interventional clinical trial within 28 days prior to the day of enrollment
* Is an immediate family member or household member of trial personnel

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Frequency of Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 175 (7 days following last dose administration)
Frequency of Unsolicited Adverse Events (AEs) | Up to Day 196 (28 days following last dose administration)
Frequency of Medically-Attended Adverse Events (MAAEs) | Up to Day 336 (6 months following last dose administration)
Frequency of Serious Adverse Events (SAEs) | Up to Day 504 (1 year following last dose administration)
Change from Baseline in Geometric Mean Titer (GMT) of Serum Neutralizing Anti-CMV Antibodies Against Epithelial Cell Infection and Against Fibroblast Infection | Baseline, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Proportion of Participants with ≥2-Fold, 3-Fold, and 4-Fold Increases in Neutralizing Antibodies (nAb) over Baseline Against Epithelial Cell Infection and Against Fibroblast Infection | Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, and Day 504

SECONDARY OUTCOMES:
Change from Baseline in GMT of Anti-Glycoprotein B (gB) Specific Immunoglobulin G (IgG) and Anti-Pentamer Specific IgG as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) of Post-Baseline/Baseline Titers | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Change from Baseline in Associated GMR of Anti-gB Specific IgG and Anti-Pentamer Specific IgG as Measured by ELISA of Post-Baseline/Baseline Titers | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Change from Baseline in GMT of Serum nAb Against Epithelial Cell Infection and Against Fibroblast Infection at Each Timepoint, in the CMV-Seropositive Group and in the CMV-Seronegative Group | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Change from Baseline in GMR of Serum nAb Against Epithelial Cell Infection and Against Fibroblast Infection at Each Timepoint, in the CMV-Seropositive Group and in the CMV-Seronegative Group | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Proportion of Participants with ≥2-Fold, 3-Fold, and 4-Fold Increases over Baseline of Serum nAb Against Epithelial Cell Infection and Against Fibroblast Infection | Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, and Day 504
Change from Baseline in GMT of Antigen-Specific IgG (ELISA) at each Timepoint in the CMV-Seropositive and CMV-Seronegative Groups | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504
Change from Baseline in GMR of Antigen-Specific IgG (ELISA) at each Timepoint in the CMV-Seropositive and CMV-Seronegative Groups | Baseline, Day 1, Day 29, Day 56, Day 84, Day 168, Day 196, Day 336, Day 504

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Benchmark Research, Sacramento, California
  - Optimal Research, Peoria, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Alliance for Multispecialty Research, Lexington, Kentucky
  - Aventiv Research Inc, Columbus, Ohio
  - Tekton Research Inc, Austin, Texas
  - Crossroads Clinical Research, Victoria, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - Foothill Family Clinic-South Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galiza EP, Khalil A, Heath PT. Update on Vaccines in Antenatal Care. Pediatr Infect Dis J. 2024 Feb 1;43(2):e60-e62. doi: 10.1097/INF.0000000000004183. Epub 2023 Dec 27. No abstract available. PMID 38190492